CLINICAL TRIAL: NCT07326007
Title: Verbal Analgesia Versus Standard Technique for Pain Control During Copper T380A Intrauterine Device Insertion in Women With Previous Cesarean Delivery: An Open-Label Randomized Controlled Trial
Brief Title: Verbal Analgesia Versus Standard Technique for Pain Control During Copper T380A Intrauterine Device Insertion in Women With Previous Cesarean Delivery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: verbal analgesia IUD-1
Record Dates: First submitted 2025-09-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verbal Analgesia (Experimental): Participants randomized to the verbal analgesia group will receive a structured communication protocol delivered by the provider throughout the IUD insertion procedure.participants will receive a structured verbal analgesia technique delivered by the provider throughout the IUD insertion procedure. The method involves using a calm, low-volume voice with steady pitch and a slow rate of speech, maintaining a non-rushed and empathetic manner intended to reduce patient anxiety and modulate pain perception. The communication is scripted to ensure consistency. Before beginning, the provider reassures the patient by saying: "You are safe here; I will guide you through every step. Please take slow, deep breaths with me." During speculum insertion, the provider continues: "You may feel some pressure now; that's normal. Keep breathing slowly." At the time of tenaculum application, the patient is prepared with: "You will feel a pinch on the cervix; it may be uncomfortable, but it will pass quick
  Interventions: Behavioral: Verbal Analgesia
- Control - Standard Technique (Active Comparator): Providers will use a standardized neutral script with brief instructions only (e.g., "I am now placing the speculum," "I am sounding the uterus," "The IUD is being inserted," "The procedure is complete"), delivered without reassurance or supportive phrasing
  Interventions: Behavioral: Providers will use a standardized neutral script with brief instructions only (e.g., "I am now placing the speculum," "I am sounding the uterus," "The IUD is being inserted," "The procedure is complet

INTERVENTIONS:
Behavioral: Verbal Analgesia — Participants randomized to the verbal analgesia group will receive a structured communication protocol delivered by the provider throughout the IUD insertion procedure.participants will receive a structured verbal analgesia technique delivered by the provider throughout the IUD insertion procedure. The method involves using a calm, low-volume voice with steady pitch and a slow rate of speech, maintaining a non-rushed and empathetic manner intended to reduce patient anxiety and modulate pain perception. The communication is scripted to ensure consistency. Before beginning, the provider reassures the patient by saying: "You are safe here; I will guide you through every step. Please take slow, deep breaths with me." During speculum insertion, the provider continues: "You may feel some pressure now; that's normal. Keep breathing slowly." At the time of tenaculum application, the patient is prepared with: "You will feel a pinch on the cervix; it may be uncomfortable, but it will pass quickl
  Arms: Verbal Analgesia
Behavioral: Providers will use a standardized neutral script with brief instructions only (e.g., "I am now placing the speculum," "I am sounding the uterus," "The IUD is being inserted," "The procedure is complet — Providers will use a standardized neutral script with brief instructions only (e.g., "I am now placing the speculum," "I am sounding the uterus," "The IUD is being inserted," "The procedure is complete"), delivered without reassurance or supportive phrasing
  Arms: Control - Standard Technique

SUMMARY:
Insertion of copper IUDs is often associated with moderate pain, which may reduce acceptance and continuation rates. Factors such as nulliparity and absence of prior vaginal delivery are known to increase pain perception. Women who have delivered only by cesarean section represent a special subgroup because their cervix has not undergone vaginal dilation and cervical remodeling, making insertion technically more difficult and often more painful. This group has been underrepresented in prior analgesia trials, highlighting an important evidence gap.

DETAILED DESCRIPTION:
Insertion of copper IUDs is often associated with moderate pain, which may reduce acceptance and continuation rates. Factors such as nulliparity and absence of prior vaginal delivery are known to increase pain perception. Women who have delivered only by cesarean section represent a special subgroup because their cervix has not undergone vaginal dilation and cervical remodeling, making insertion technically more difficult and often more painful. This group has been underrepresented in prior analgesia trials, highlighting an important evidence gap.

Pharmacological interventions (NSAIDs, opioids, local anesthetics) have shown inconsistent results. A randomized controlled trial demonstrated that verbal analgesia, using calm voice, reassurance, and continuous communication, was as effective as tramadol for IUD insertion among nulliparous women. To date, no randomized study has specifically addressed women delivered only by cesarean section

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years.

  * Desire for Copper T380A IUD.
  * Delivery history limited to cesarean section(s), no vaginal delivery

Exclusion Criteria:

* o Current pelvic infection, cervicitis, or vaginitis.

  * Uterine anomalies or fibroids distorting the cavity.
  * Contraindication to copper IUD procedure, and use of any analgesic medication within the last 6-8 hours prior to insertion.
  * Pregnancy or suspected pregnancy.
  * Severe dysmenorrhea requiring narcotics

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
pain during IUD insertion | immediately after IUD insertion. at the time if IUD release into the uterine cavity
  Pain intensity measured by a 0-10 Numerical Rating Scale (NRS) immediately after IUD release in the uterine cavity, where 0 = "no pain" and 10 = "worst pain imaginable

SECONDARY OUTCOMES:
Clinician-rated ease of insertion | Immediately after completion of IUD insertion procedure
  It will be measured by a 0-10 NRS-like scale immediately after the procedure, where 0 = very easy insertion and 10 = most difficult insertion.
Patient satisfaction | at the end of procedure before discharge from clinic
  It will be measured usinga 0-10 NRS-like scale at the end of the visit, where 0 = no satisfaction and 10 = maximum satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Al Gezeera Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided